CLINICAL TRIAL: NCT05559190
Title: Effect of Preoperative Pulsed Electromagnetic Field and Abdominal Exercises on Muscle Strength Post Ventral Hernioplasty
Brief Title: Effect of a Preoperative Pulsed Electromagnetic Field and Abdominal Exercises on Muscle Strength Post Ventral Hernioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohamed Ahmed Elsayeh, Lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002965
Record Dates: First submitted 2022-09-24; First posted 2022-09-29 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Hernia, Ventral
Keywords: pulsed electromagnetic field; abdominal exercises; ventral hernia repair
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pulsed electromagnetic field and selected graduated abdominal exercises (group A) (Experimental): The interventions were done preoperatively, received pulsed electromagnetic therapy (PEMFT) on abdominal muscles,15 Hz frequency, 20 gauss amplitude with a rectangular waveform, for 20 minutes then they performed the selected graduated abdominal strengthening exercises for 30 minutes, three sessions per week for six weeks.
  Interventions: Other: Pulsed electromagnetic field; Other: Graduated abdominal strengthening exercises
- Selected graduated abdominal exercises (group B) (Active Comparator): The interventions were done preoperatively, patients performed the selected graduated abdominal strengthening exercises for 30 minutes, three sessions per week for six weeks.
  Interventions: Other: Graduated abdominal strengthening exercises
- Pulsed electromagnetic field (group C) (Active Comparator): The interventions were done preoperatively, they received pulsed electromagnetic therapy (PEMFT) on abdominal muscles,15 Hz frequency, 20 gauss amplitude with a rectangular waveform, for 20 minutes only.
  Interventions: Other: Pulsed electromagnetic field
- Control group (No Intervention): Patients were instructed to presume in normal activities of daily living preoperatively, without any abdominal exercises or PEMFT.

INTERVENTIONS:
Other: Pulsed electromagnetic field — Pulsed electromagnetic field therapy was applied directly over the abdominal muscle from a supine position after the removal of metals or things that can be affected by a magnetic field will be assured prior to magnetic field application. The treatment parameters were set as 15 Hz frequency, 20 gauss amplitude with a rectangular waveform for 20 minutes.
  Arms: Pulsed electromagnetic field (group C); Pulsed electromagnetic field and selected graduated abdominal exercises (group A)
Other: Graduated abdominal strengthening exercises — Four specific muscle core exercises were performed
  Arms: Pulsed electromagnetic field and selected graduated abdominal exercises (group A); Selected graduated abdominal exercises (group B)

SUMMARY:
The aim of this study is to investigate the impact of a preoperative pulsed electromagnetic field and abdominal exercises on muscle strength post ventral hernioplasty.

DETAILED DESCRIPTION:
Sixty patients, 25-40 years old, diagnosed with a ventral hernia and consulted for surgical hernia repair, preoperatively, were randomly assigned either into pulsed electromagnetic therapy and graduated abdominal strengthening exercises group (group A), graduated abdominal strengthening exercises group (group B), pulsed electromagnetic therapy group (group C) or group D who is instructed to presume in normal activities of daily living preoperatively, without any abdominal exercises or PEMF. All treatment interventions were applied at a frequency of three sessions per week for six weeks preoperatively. Abdominal muscle torque was measured by a biodex isokinetic dynamometer preoperatively at baseline and after six weeks of intervention and after four months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Being subjects of both genders.
* Between the age of 25-40 years.
* Diagnosed with a ventral hernia (Grade II & III) based on surgeon assessment and desired an elective surgical repair.
* Able to act in the abdominal training program.

Exclusion Criteria:

* Patients with a strangulated hernia.
* Bowel obstruction, peritonitis or perforation.
* Urgent surgery indication.
* Less than one-year abdominal surgery.
* Infection (local or systemic).
* Orthopedic problem, or neurological impairment that interfere with patient ability to act in the abdominal training program.
* Pregnant women.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
the change in the abdominal muscle torque | Baseline and six weeks after the intervention preoperatively and after four weeks postoperative as follow up
  measured by biodex isokinetic

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa MA Elsayeh, PhD, Principal Investigator — Lecturer at Faculty of Physical Therapy, Cairo University
Locations (1):
- Shaimaa Mohamed Ahmed Elsayeh, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No